CLINICAL TRIAL: NCT02268968
Title: Use of Topical Lidocaine to Reduce Pain in Preterm Infants Receiving Nasal Contiuous Positive Airway Pressure
Brief Title: Use of Topical Lidocaine to Reduce Pain in Preterm Infants Receiving Nasal CPAP Continuous Positive Airway Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdel-Hady, Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS 012
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Other Preterm Infants
Keywords: Topical Lidocaine; Nasal CPAP; Pain; Preterm Infants; Salivary cortisol
MeSH Terms: conditions — Pain | interventions — Lidocaine; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental): Intervention: Topical lidocaine gel 2% (0.3 ml/kg) will be applied once only to the nostrils and nasal CPAP prong 5 minutes prior to the application of nasal CPAP
  Interventions: Drug: Lidocaine 2% Gel
- Control (No Intervention): No topical lidocaine will be used prior to application of nasal CPAP

INTERVENTIONS:
Drug: Lidocaine 2% Gel — Lidocaine 2% gel will be applied to nostrils and nasal CPAP prong 5 minutes prior to application of nasal CPAP
  Other Names: Xylocaine jelly 2%
  Arms: Lidocaine

SUMMARY:
The main purpose of this study is to evaluate the relative efficacy of topical lidocaine on reducing pain associated with the application of nasal CPAP in preterm infants

DETAILED DESCRIPTION:
Preterm infants admitted to NICUs are exposed to a range of painful procedures. The exposure to pain during this critical of brain development may have adverse consequences. Application of nasal CPAP is one of the painful procedures. A consensus statement on neonatal pain made recommendations for analgesia for neonatal procedures. Topical lidocaine is frequently used as a topical anesthetic during venipuncture, heel lancing, circumcision, endotracheal intubations, nasogastric tube insertion, endoscopy and bronchoscopy. However, the use of topical lidocaine for its analgesic effect on application of nasal CPAP has not been evaluated.

This study proposes a randomized controlled trial to evaluate the relative efficacy of topical lidocaine on reducing pain associated with the application of nasal CPAP in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants < 37 weeks gestation
* Admitted to NICU, Mansoura University Children's Hospital
* Respiratory distress requiring use of nasal CPAP
* Informed consent obtained

Exclusion Criteria:

* Serious, life-threatening malformations
* Use of sedation, analgesia in the preceding 72 hours
* Those who undergo any surgical intervention
* Those who undergo any painful procedures as venipuncture, intubation, suctioning, blood sampling, heel-prick, catheterization 30 minutes before assessment
* Those with signs of nasal injuries at the time of application of nCPAP
* Necrotizing enterocolitis

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The Premature Infant Pain (PIPP) Scale | Immediately after application of nasal CPAP (approx 5 min)
  PIPP comprises 3 behavioral variables (time of brow bulge, eye squeeze, and naso-labial furrow), 2 physiologic variables (changes in heart rate and SpO2), and 2 contextual variables (gestational age and behavioral state). Behavioral state ranges from "active/awake, eyes open, facial movements" to "quiet/sleep, eyes closed, no facial movements." Every variable will be scored on a scale from 0 to 3. A total score the sum of total of points indicating: lack of pain (0-6), mild -moderate pain (6-12) and severe pain (above 12). PIPP has documented reliability and validity and have been used previously in several studies in neonates. PIPP score measurement will be based on video recording the infant for 45 seconds. Three different DVDs will be compiled with the sets in random order. Three different nurses from NICU will be recruited to evaluate the segments. They will not be informed of the nature of the study. All 3 nurses are trained in performing the PIPP.

SECONDARY OUTCOMES:
Salivary cortisol | 30 minute after application of nasal CPAP
  Salivary samples will be obtained 30 minutes after application of nasal CPAP using sterile single channel 500 μl pipette (Dragon Laboratory Instruments Limited, Beijing 101318 China). After collection, the saliva wll be centrifuged, frozen and stored at -70°C. The samples will later analysed using ELISA technique; IBL kits (IBL International GmbH, Flughafenstr. 52A, 22335 Hamburg, Germany).
Duration of first cry | Immediately after application of nasal CPAP (approx 5 min)
  The duration of the first cry will be defined as audible distressed vocalizations with a continuous pattern before a quiet interval of 5 seconds soon after application of nasal CPAP
Possible adverse effects to lidocaine | Within 72 hours of application of topical lidocaine gel
  CNS side effects as irritability, nervousness, confusion, vomiting, twitching, tremors, convulsions, unconsciousness, respiratory depression, and arrest.
  Cardiovascular side effects: bradycardia, hypotension, and cardiovascular collapse, and cardiac arrest.
  Allergic: urticaria, edema, or anaphylactic reactions
Nasal trauma | 24 hours after application of nasal CPAP
  The nose of enrolled infants will be assessed for any sign of injury 24 hours after application of nasal CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Hesham E Abdel-Hady, MD, PhD, Principal Investigator — Mansoura University Children Hospital
Locations (1):
- Neonatal Intensive Care Unit, Mansoura University Children Hospital, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Britto CD, Rao Pn S, Nesargi S, Nair S, Rao S, Thilagavathy T, Ramesh A, Bhat S. PAIN--perception and assessment of painful procedures in the NICU. J Trop Pediatr. 2014 Dec;60(6):422-7. doi: 10.1093/tropej/fmu039. Epub 2014 Jul 21. PMID 25053125
- [Background] Prevention and management of pain and stress in the neonate. American Academy of Pediatrics. Committee on Fetus and Newborn. Committee on Drugs. Section on Anesthesiology. Section on Surgery. Canadian Paediatric Society. Fetus and Newborn Committee. Pediatrics. 2000 Feb;105(2):454-61. PMID 10654977
- [Background] Bendixen D, Halvorsen AC, Hjelt K, Flachs H. Lignocaine gel used for lubrication of intranasal and endotracheal tubes in premature neonates. Acta Paediatr. 1994 May;83(5):493-7. doi: 10.1111/j.1651-2227.1994.tb13065.x. PMID 8086725
- [Background] Lillieborg S, Otterbom I, Ahlen K. Topical anaesthesia in neonates, infants and children. Br J Anaesth. 2004 Mar;92(3):450; author reply 450-1. doi: 10.1093/bja/aeh522. No abstract available. PMID 14970141